CLINICAL TRIAL: NCT02443311
Title: A Comparative Clinical and Immunohistochemical Study Between Topical Pimecrolimus and Corticosteroid in Treatment of Oral Lichen Planus
Brief Title: Clinical and Immunohistochemical Effect of Topical Pimecrolimus in Treatment of Oral Lichen Planus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ola Mohamed Ezzatt, Lecturer of oral medicine and periodontology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-RECD 1214401
Record Dates: First submitted 2015-05-10; First posted 2015-05-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — pimecrolimus; Betamethasone Valerate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Experimental): Pimecrolimus 1% cream (Elidel, Novartis Pharmaceuticals, East Hanover, NJ)+ custom made hydrophilic Adhesive gel base (Department of Pharmaceutics and Industrial Pharmacy. Faculty of Pharmacy. Ain Shams University) 4 Times/day for 4 weeks
  Interventions: Drug: Pimecrolimus 1% cream
- Group II (Active Comparator): Betamethasone 17-valerate 0.1% cream (Betnovate, GlaxoSmithKline, Cairo, Egypt)+ custom made hydrophilic Adhesive gel base (Department of Pharmaceutics and Industrial Pharmacy. Faculty of Pharmacy. Ain Shams University) 4 Times/day for 4 weeks
  Interventions: Drug: Betamethasone 17-valerate 0.1% cream

INTERVENTIONS:
Drug: Pimecrolimus 1% cream — Patients were instructed to apply a thin layer of mixed equal amounts (½ ml) of the study medication and the adhesive gel base per application guided by the graduation on the plastic syringe on the oral lesions, 4 times daily, for a total of 1month. The patients were asked not to eat, drink, for 30 minutes after each application.
  Arms: Group I
Drug: Betamethasone 17-valerate 0.1% cream — Patients were instructed to apply a thin layer of mixed equal amounts (½ ml) of the study medication and the adhesive gel base per application guided by the graduation on the plastic syringe on the oral lesions, 4 times daily, for a total of 1month. The patients were asked not to eat, drink, for 30 minutes after each application.Topical antifungal Miconazole 2% gel (Miconaz, oral Medical Union Pharmaceutical, Cairo, Egypt) was applied only in the fourth week of treatment period to avoid secondary candidiosis
  Arms: Group II

SUMMARY:
Oral lichen planus (OLP) is a chronic disease characterized by periods of remission and relapse. Therapeutic objectives for OLP should be to quickly reduce disease symptoms by targeting pathophysiological pathways, and to provide long-term management by reducing recurrences. Pimecrolimus is a novel topical selective inflammatory cytokine release inhibitor; considering its mechanism of action it is reasonable to theorize that pimecrolimus may effectively treat OLP without the potential side effects that are associated with corticosteroids.

DETAILED DESCRIPTION:
Lichen planus is a chronic, immunological, mucocutaneous disease, characterized by periods of remission and relapse1. Oral lichen planus (OLP) is one of the most common mucocutaneous diseases manifesting in the oral cavity, and the oral mucosa may be the only site of involvement 2, with variable incidence between 0.5% and 4% 3. Three major clinical forms of OLP (reticular, erosive/ ulcerative, and erythematous/atrophic) have been recognized, which could alternate and overlap in a dynamic state as disease progresses. Ulceration is the most severe form that it interferes with eating, speech, and swallowing. Erosive OLP lasts for years, resistance to treatment and spontaneous remissions are rare 4,5. Oral lichen planus is a T-cell-mediated chronic inflammatory oral mucosal disease. Both antigen-specific and non-specific mechanisms may be involved in the pathogenesis of OLP. Antigen-specific mechanisms include antigen presentation by basal keratinocytes to CD4+ helper T-cells that are stimulated to secrete the T helper -1 cytokines IL-2 and IFN-γ. Subsequently, CD8+ cytotoxic T-cells may be activated which then trigger basal keratinocyte apoptosis in OLP. While, non-specific mechanisms include mast cell degranulation and matrix metalloproteinase (MMP) activation in OLP lesions 6. The best known treatment of OLP remains high-potency topical corticosteroids7. However, corticosteroids are known to induce local atrophy, fragility, and telangiectasias, and to promote infections, including acute candidiasis. They also have theoretical risks of lowering local immunity, corticosteroids can exert their effects on the immune system by modulating transcription of genes in cells involved in immune response and other cell types; therefore this mode of action is not selective for the pathogenesis of lichen planus 8-10. A recent Cochrane review showed only little evidence for superiority of the assessed interventions over placebo for palliation of symptomatic OLP and recommended the need of randomized clinical trials on new therapies 11. Pimecrolimus a novel topical selective inflammatory cytokine release inhibitor; that binds to intra-cytoplsmic protein (macrophillin-12) subsequently inhibiting dephosphorylation of nuclear factor of activated T cells by calcineurin; this markedly reduces T-cell cytokine production. Given the T-cell-mediated pathogenesis of OLP, application of this calcineurin inhibitor seems to be a promising therapeutic option 12-14. Several case studies and open-label trials used topical pimecrolimus in treatment of OLP reported beneficial effects 12,15. Few prospective, randomized, vehicle-controlled studies have also been conducted and proved benefit of pimecrolimus over placebo 16,10,17. And one recent prospective study compared the effect of topical pimecrolimus with topical corticosteroid in treatment of OLP 18. The purpose of this study was to compare the effectiveness of topical pimecrolimus 1% with topical corticosteroid, in the treatment of oral erosive and atrophic lichen planus as a prospective, comparative clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* clinically and histologically confirmed painful Erosive or Atrophic OLP
* free from any systemic diseases using medical questionnaire guided by Cornell Medical Index

Exclusion Criteria:

* history of drug induced lichenoid lesions
* potential treatment of OLP for less than 2 weeks by topical and 4 weeks systemic therapy before study start
* pregnant or breast-feeding women,
* smoking and
* known hypersensitivity or severe adverse effects to the treatment drugs or to any ingredient of their preparation
* loss of paliability or flexibility in the tissues involved by the oral lesions or histological signs of epithelial dysplasia or lichenoid lesions within the biopsied sites.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-09; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
clinical scoring (CS) | 2 months/ once per week for one months then after 2 months
  0 represented no lesion/normal mucosa; 1, mild white striae/no erythematous area; 2, white striae with atrophic area less than 1 cm²; 3, white striae with atrophic area more than 1 cm²; 4, white striae with erosive area less than 1 4 cm²; and 5, white striae with erosive area more than 1 cm²
visual analog scale (VAS) | 2 months/ once per week for one months then after 2 months
  Patients also ranked the severity of pain and burning sensation on 100-mm visual analog scale

SECONDARY OUTCOMES:
CD4+,CD8+, CD133 | baseline and after 1 month treatment
  Immunohistochemical analysis